CLINICAL TRIAL: NCT04632173
Title: HERODOTUS: Head and Neck cancERs International cOviD-19 collabOraTion
Brief Title: Head and Neck cancERs International cOviD-19 collabOraTion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hellenic Cooperative Oncology Group (Other)
Collaborators: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Grupo Español de Tratamiento de Tumores de Cabeza y Cuello (Other); National Cancer Centre, Singapore (Other); Emory University (Other); University of Toronto (Other); University of Birmingham (Other); The University of Queensland (Other)
Responsible Party: Principal Investigator, Amanda Psyrri, Associate Professor of Medical Oncology, Hellenic Cooperative Oncology Group
Other Study IDs: HERODOTUS
Record Dates: First submitted 2020-11-15; First posted 2020-11-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Head and Neck Cancer; Covid19
MeSH Terms: conditions — Head and Neck Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non interventional study — There is no intervention

SUMMARY:
To develop an International registry on head and neck cancer patients infected with COVID-19

DETAILED DESCRIPTION:
On 11 March, the World Health Organization (WHO) formally declared the corona virus disease-19 (COVID-19) outbreak a pandemic. After the first cluster of cases emerged from Wuhan, in China, at the end of 2019, up today almost 2 million cases of infections from severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) have been diagnosed across all five continents in the last few months.By the end of February 2020 COVID-19 had already hit Europe hard, particularly Italy, with 12462 confirmed cases according to the Istituto Superiore di Sanità as of March 11th, and 827 deaths. Considering the high transmissibility and the severe disease occurrence in a fraction of the population, healthcare systems face a great challenge. The estimated risk of death varies, indeed from the 12% In China at the peak of the epidemic, to ≈1% in less affected regions including Europe, USA, Australia, Latin America, Iran, and Canada.COVID-19 morbidity and mortality have been linked to elderly age and comorbidities, leading to a poorer outcome from the viral infection in frail patients, more often resulting in hospitalization, intensive care unit admittance and need for invasive tracheal intubation. Among 2 such individuals, cancer patients represent a large subgroup at high risk of developing coronavirus infection and its severe complications. A recent nationwide analysis in China demonstrated that, of 1590 COVID-19 cases from 575 hospitals, 18 had a history of cancer (1% vs 0.29% of cancer incidence in the overall Chinese population, respectively), with lung cancer as the most frequent diagnosis. Patients with cancer were observed to have a higher risk of severe events compared with patients without cancer (39 vs 8%; p = 0.0003). Moreover, cancer patients who underwent recent chemotherapy or surgery had a higher risk of clinically severe events than did those not receive treatment. With the limit of a small sample size, the authors concluded that patients with cancer might have a higher risk of COVID-19, and poorer outcomes, than individuals without cancer. As a consequence, they recommended considering an intentional postponement of adjuvant chemotherapy or elective surgery for stable cancer in endemic areas. Nevertheless, as subsequently highlighted by other authors, the true incidence of COVID-19 in patients with cancer would be more informative in assessing whether such patients have an increased risk (and morbidity) from this viral illness. Furthermore, COVID-19 pandemic has led to delay in cancer diagnosis and modifications in cancer treatment to limit as much as possible the number of patients in order to reduce the risks of contamination by the SARS-Cov-2 virus for both patients and the caregivers. Arduino PG et al reported a substantial delay in oral cancer diagnosis in north-west Italy due to COVID19 outbreak. In addition, the management of cancer patients is modified during the COVID-19 pandemic including delays in surgery, delays and modification of radiation treatment schedule. Cancer Societies have issued treatment guidelines of cancer patients during COVID-19 which include treatment adjustments the impact of which is currently unknown. In addition, the coexistence of COVID-19 and cancer may increase the incidence of treatment complications such as postoperative thrombosis and pulmonary emboli. For COVID-19 + thyroid cancer patients treated with tyrosine kinase inhibitors, treatment complications and outcomes are very relevant clinical questions. Furthermore, the limited cancer patient population described in this first report from the literature, was characterized by the lack of individuals receiving anticancer immunotherapy. Indeed, only chemotherapy and surgery were cited among treatments received by patients in the month prior to developing COVID-19. Maybe, this could simply be due to the casualty of a small sample, or otherwise, it could suggest that cancer patients receiving immunotherapy are less prone to develop COVID-19 or to be admitted in hospital due to severe coronavirus symptoms. Currently, we are aware of the probably higher incidence of misdiagnosed coronavirus infections compared with that reported and updated every day; it is likely that a large portion of healthy and young population develop COVID-19 with mild symptoms, not requiring hospital admittance and thus escaping the laboratory confirmation of the disease.

Cancer patients undergoing treatment with anti-PD-1/PD-L1 currently used in everyday practice to treat head and neck carcinoma constitute a growing oncological population. Their specific susceptibility to bacterial or viral infections has not been investigated. Considering that immunotherapy with Immune Checkpoint Inhibitors (ICI) is able to restore the cellular immunocompetence, as it was previously suggested in the context of influenza infection, the patient undergoing immune checkpoint blockade could be more immunocompetent than cancer patients undergoing chemotherapy. In the recent weeks, in the countries heavily affected by the COVID-19 outbreak, such as Italy, scientific associations recommended the prudential postponing of active cancer treatments,especially for stable patients not needing urgent interventions. On one hand, this recommendation could be reasonable for advanced cancer patients receiving chemotherapy, with the risk of hematological toxicity and of worsening an immunosuppressed status, thus favoring COVID-19 morbidity. On the other hand, some oncologists are even currently wondering about the risk of administering ICI in the middle of the COVID-19 outbreak, essentially due to two major concerns.

The first seems to be represented by the potential overlap between the coronavirus-related interstitial pneumonia and the possible pneumological toxicity from anti-PD-1/PD-L1 agents.

Even if lung toxicity is not the most frequent adverse event of ICI, it can be life threatening.

The overall incidence rate of ICI-related pneumonitis ranges from 2.5-5% with anti-PD1/PDL1 monotherapy to 7-10% with anti-CTLA-4/anti-PD-1 combination therapy. The dominant radiological pattern of lung Immune-related Adverse Events (irAEs) is organizing pneumonia,but ICI-related pneumonitis could exhibit a variety of patterns, also including nonspecific interstitial pneumonitis. Despite being rarer than other irAEs, pneumonitis is the most fatal Adverse Event (AE) associated with PD-1/PD-L1 inhibitor therapy, accounting for 35% of treatment-related toxic deaths. Considering that underlying lung disease, particularly including interstitial pneumopathy, is considered a risk factor for ICI-related pneumonitis, it could be reasonable taking into account the risk of treating patients while they are developing an initial form of COVID-19. The synergy between the two lung injuries, despite only hypothetical, cannot be surely ruled out. Nevertheless, such an epidemiological coincidence should not prevent the oncologist from offering a potentially effective and often well-tolerated treatment even in the middle of the COVID-19 outbreak, since the duration of the pandemic is still currently unpredictable. The second concern seems to be represented by a possible negative interference of ICI in the pathogenesis of COVID-19. Cytokine-release syndrome (CRS) is a phenomenon of immune hyperactivation typically described in the setting of T cell-engaging immunotherapy, including Chimeric Antigen Receptor (CAR)-T cell therapy but also anti-PD-1 agents. CRS is characterized by elevated levels of Interleukin (IL)-6, Interferon (IFN)- γ and other cytokines, provoking consequences and symptoms related to immune activation, ranging from fever, malaise and myalgias to severe organ toxicity, lung failure and death. In parallel, one of the most important mechanisms underlying the deterioration of disease in COVID-19 is represented by the cytokine storm, leading to acute respiratory distress syndrome or even multiple organ failure. The cytometric analyses of COVID-19 patients showed reduced counts of peripheral CD4 and CD8 T cells, while their status was hyperactivated. In addition, an increased concentration of highly proinflammatory CCR6+ Th17 in CD4 T cells has been reported, and CD8 T cells were found to harbor high concentrations of cytotoxic granules, suggesting that over activation of T cells tends to contribute to the severe immune injury of the disease. Moreover, the pathological findings associated with acute respiratory distress syndrome in COVID-19 showed abundant interstitial mononuclear inflammatory infiltrate in the lungs, dominated by lymphocytes, once again implying that the immune hyperactivation mechanisms are at least partially accountable for COVID-19 severity. Considering these aspects, the hypothesis of a synergy between ICI mechanisms and COVID-19 pathogenesis, both contributing to a counter-producing immune hyperactivation, cannot be excluded. In spite of this fascinating rationale, we should remember that ICI-induced CRS is a quite rare phenomenon as well as that the cytokine storm is not an early event in the COVID-19 pathogenesis, indeed characterizing the late phase of its most severe manifestation, occurring in a minority of patients. It is not likely that cancer patients are still receiving ICI during this phase of the viral illness. Obviously, in the current pandemic scenario, careful attention should be dedicated in delaying treatment for those patients presenting flu-like symptoms at the time of the intended ICI treatment.

Considering this background, we propose a global registry to describe and monitor head and neck cancer patients with COVID-19; identify factor associated with severe complications; develop a tailored risk assessment strategy for head and neck cancer patients; and develop treatment recommendations for head and neck cancer patients.

ELIGIBILITY:
Inclusion Criteria:

Any head and neck cancer patients (including salivary gland, thyroid, nasal and paranasal cancer with a COVID-19 diagnosis defined as any of the following:

* Laboratory confirmed [Real Time - Polymerase Chain Reaction (RT-PCR) technique] COVID-19.
* Suspected COVID-19 cases; diagnosed clinically based on symptoms (fever >37.5°, decrease of oximeter saturation of at least 5 %, cough, diarrhoea, otitis, dysgeusia, anosmia, myalgia, arthralgia, conjunctivitis and rhinorrhea and exposure to confirmed COVID-19 positive case (laboratory confirmation).
* Clinically diagnosed cases; suspected cases with lung imaging features consistent with coronavirus pneumonia.
* Asymptomatic cases; diagnosed based on positive viral nucleic acid test results but without any COVID- 19 symptoms

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a longitudinal multi-centre study on head and neck cancer patients (any age, sex, histology, stage, in active treatment as well as in clinical follow-up) who contract COVID-19.
  Information on clinical features, clinical course, management and outcomes will be collected for both, head and neck cancers and COVID-19 infection. Considering the limited data available about COVID-19 evolution, the sample size will be not anticipated. However, with about 150 centers and a median of 5 patients at every center, a sample size of 750 patients approximately can produce a confidence interval for the categorical estimate of +/-2%. Clinical data will be extracted from medical records of consecutive patients from November 1st, 2019 until January 31 2021.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Demographic features | Nov 1 2019 to January 31 2021
  age, performance status etc
prevalence of comorbidities in head and neck cancer patients with COVID-19 | Nov 1 2019 to January 31 2021
proportion of head and neck cancer patients experiencing severe adverse events | Nov 1 2019 to January 31 2021
proportion of head and neck cancer patients by COVID-19 clinical course severity | Nov 1 2019 to January 31 2021
proportion of head and neck cancer patients with COVID-19 who received chemotherapy, surgery, radiotherapy, immune check point inhibitors in the last 3 months before, as well as during, COVID-19 infection | Nov 1 2019 to January 31 2021
predictive factors of severe adverse events in head and neck cancer patients with COVID-19 including cancer-related treatment | Nov 1 2019 to January 31 2021
prognostic factors of head and neck cancer patients with COVID-19 including cancer related treatment including Human papilloma virus(HPV). | Nov 1 2019 to January 31 2021

CONTACTS AND LOCATIONS:
Overall Officials: Evita Fragou, Study Director — HeCOG
Locations (3):
- "Attikon" University Hospital, Chaïdári, Athens, Greece
- Lisa Licitra, Milan, Italy
- National Cancer Centre (NCC)- Radiation Oncology Dept, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No